CLINICAL TRIAL: NCT00001805
Title: A Phase II Clinical Trial of Suppression of Human Antimouse Antibody and Human Antitoxin Response to Immunotoxin LMB-1 by Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990071; 99-C-0071
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms
Keywords: Breast Cancer; Colon Cancer; Gastric Cancer; Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This is a phase II clinical and pharmacokinetic study of suppression of human antimouse (HAMA) and antitoxin antibodies (HATA) to immunotoxin LMB-1 by Rituximab (anti-CD20). The primary objective of this study is to determine the effect of Rituximab on HAMA and HATA response to LMB-1 administered to patients with advanced carcinoma that express the B3 antigen. Other objectives include evaluation of the pharmacokinetics and anti-tumor effects.

DETAILED DESCRIPTION:
This is a phase II clinical and pharmacokinetic study of suppression of human antimouse (HAMA) and antitoxin antibodies (HATA) to immunotoxin LMB-1 by Rituximab (anti-CD20). The primary objective of this study is to determine the effect of Rituximab on HAMA and HATA response to LMB-1 administered to patients with advanced carcinoma that express the B3 antigen. Other objectives include evaluation of the pharmacokinetics and anti-tumor effects.

ELIGIBILITY:
Patients must have advanced stage solid tumor with histologically or cytologically proven evaluable or measurable disease and who are refractory to standard treatment for their malignancy or for whom no effective standard therapy exists.

Must have the presence of B3 antigen on the surface of greater than 30% of the tumor cells.

Must be greater than or equal to 18 years old and be able to give informed consent.

Must have an ECOG performance status of 0 or 1 and a minimum life expectancy of 3 months.

Must have normal renal function (Creatinine less than or equal to 1.4 mg/dl), SGOT and SGPT less than or equal to 2.5 x of the upper limits of normal. Total bilirubin less than 1.5 mg/dL; AGC greater than or equal to 1.5 x 10(3) microliter; platelets greater than 100,000 per mm(3).

Must have recovered from the toxic effects of prior chemotherapy or radiation therapy. At least 3 weeks must have elapsed since the last dose of chemotherapy, hormonal therapy or radiation therapy. At least six weeks must have elapsed since the last dose of Mitomycin C and a nitrosourea.

Must not have serum neutralizing antibodies to LMB-1.

Must not have positive hepatitis B surface antigen, hepatitis C antibody or HIV.

Must not have a history of coronary artery disease, NY class II-IV CHF, arrhythmia requiring treatment and any contraindication to pressor therapy.

Must not have FEV1 and FVC less than or equal to 65% of the predicted value.

Must not have baseline serum albumin of less than 3.0 g/dl.

Must not have a history of CNS metastasis and/or known seizure disorders, or concurrent malignancy.

Must not have an acute bacterial infection that requires antibiotic therapy (unless infection is completely resolved).

Must not have any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.

Must not be pregnant or breastfeeding. Patients of childbearing potential must agree to use an effective method of contraception.

Must not have a history of allergic reaction to penicillin.

Must not have lymphoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1999-03; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Grossbard ML, Lambert JM, Goldmacher VS, Spector NL, Kinsella J, Eliseo L, Coral F, Taylor JA, Blattler WA, Epstein CL, et al. Anti-B4-blocked ricin: a phase I trial of 7-day continuous infusion in patients with B-cell neoplasms. J Clin Oncol. 1993 Apr;11(4):726-37. doi: 10.1200/JCO.1993.11.4.726. PMID 7683045
- [Background] Amlot PL, Stone MJ, Cunningham D, Fay J, Newman J, Collins R, May R, McCarthy M, Richardson J, Ghetie V, et al. A phase I study of an anti-CD22-deglycosylated ricin A chain immunotoxin in the treatment of B-cell lymphomas resistant to conventional therapy. Blood. 1993 Nov 1;82(9):2624-33. PMID 8219217
- [Background] Byers VS, Rodvien R, Grant K, Durrant LG, Hudson KH, Baldwin RW, Scannon PJ. Phase I study of monoclonal antibody-ricin A chain immunotoxin XomaZyme-791 in patients with metastatic colon cancer. Cancer Res. 1989 Nov 1;49(21):6153-60. PMID 2790828